CLINICAL TRIAL: NCT05361343
Title: First Line Prevent Age Study
Acronym: FLIPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prevent Age Resort "Pervaya Liniya" (Other)
Responsible Party: Principal Investigator, Anna Ratnikova, Cardiologist, MD, PhD, Chief physician, PervayaLiniyaResort, Russia, Saint Petersburg State University, Russia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FLIPS-1
Record Dates: First submitted 2022-04-15; First posted 2022-05-04 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Healthy Aging; Healthy Lifestyle; Healthy Diet
MeSH Terms: interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Other): 1. Nutrition: intermittent fasting;
  2. Physical activity: medium-intensity or high-intensity physical activity;
  3. Hypoxic training (at least three per visit to the center);
  4. correction of hygiene and sleep duration, relaxation techniques, cognitive behavioral therapy for insomnia.
  5. Individual motivational counseling.
  Interventions: Other: 1. Nutrition; 2. Physical activity; 3. Hypoxic training; 4. Menthal heals improvement

INTERVENTIONS:
Other: 1. Nutrition; 2. Physical activity; 3. Hypoxic training; 4. Menthal heals improvement — 1. Nutrition: intermittent fasting;
  2. Physical activity: medium-intensity or high-intensity physical activity;
  3. Hypoxic training (at least three per visit to the center);
  4. correction of hygiene and sleep duration, relaxation techniques, cognitive behavioral therapy for insomnia.
  5. Individual motivational counseling.

SUMMARY:
To prove the effectiveness of complex wellness programs in terms of maintaining active longevity, including motivational counseling, high-intensity training, intermittent fasting, hypoxic training, as well as practices for achieving healthy sleep and mental well-being.

Clinical-instrumental, single-centre, prospective, open-label, non-randomized, sequential enrollment study with blinded endpoint analysis

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18;
* No significant (affecting the functional state) "active" diseases: acute diseases and exacerbations of chronic diseases;
* Interest in active longevity and willingness to participate in research.
* Signed informed consent.

Exclusion Criteria:

* Age up to 18 years;
* Severe or moderate comorbidities;
* Rheumatological (systemic / autoimmune) diseases of any severity;
* Intestinal infections (within 3 months);
* SARS / pneumonia, other diseases accompanied by systemic inflammation during the last 2 months;
* Chronic inflammatory bowel disease;
* Major surgery within the last 3 months
* Intoxication (alcohol, drugs, other toxins);
* Oncological disease (except for basalioma) out of remission;
* Persons with mental illness;
* Diabetes;
* Syndrome of obstructive sleep apnea of moderate and severe severity;
* Low adherence to lifestyle interventions, including physical activity of less than 150 minutes of aerobic activity per week (at least two days per week) or 75 minutes of vigorous exercise (at least 3 days per week).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
improved endothelial function | First point: 1 week (2nd visit). Second oint after 6 - 13 months (3rd visit)
  improvement of flow-mediated vasodilatation measured by ultrasound (cuff test)
improved quality of night sleep | First point: 1 week (2nd visit). Second oint after 6 - 13 months (3rd visit)
  improvement in nighttime sleep quality assessed by a Pittsburgh Sleep Quality Scale
Reducing the degree of anxiety | First point: 1 week (2nd visit). Second oint after 6 - 13 months (3rd visit)
  Reduction in the degree of anxiety according to the assessment of the Spielberger test

SECONDARY OUTCOMES:
increased self-esteem | First point: 1 week (2nd visit). Second oint after 6 - 13 months (3rd visit)
  increasing the level of self-esteem based on the results of the analysis of the Dembo-Rubinstein questionnaire
improved quality of night sleep | First point: 1 week (2nd visit). Second oint after 6 - 13 months (3rd visit)
  improvement in nighttime sleep quality assessed by a sleep indicator scale

CONTACTS AND LOCATIONS:
Locations (1):
- First Line Health Care Resort, Saint Petersburg, Russia